CLINICAL TRIAL: NCT06445166
Title: A Multicenter Phase II Study of Propranolol for the Treatment of Kaposi Sarcoma in Adults
Brief Title: Propranolol for the Treatment of Kaposi Sarcoma in Adults
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: The Foundation for Barnes-Jewish Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202408004
Record Dates: First submitted 2024-05-31; First posted 2024-06-06 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Kaposi Sarcoma
Keywords: Propranolol; Kaposi; Sarcoma; Phase II; HIV
MeSH Terms: conditions — Sarcoma, Kaposi; Sarcoma | interventions — Propranolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Propranolol (Experimental): Begin at 1/2 the target dose for 7 days, followed by a tolerability assessment. Patients intolerant of the half dose will discontinue treatment. Patients who tolerate the 1/2 dose will increase to the full dose for 7 days, after which tolerability will be assessed on day 8. Patients who do not tolerate the full dose will taper and then discontinue treatment. Those who continue will take the target dose for 12 weeks. At week 13 time point, tolerability and response assessment will be performed:
  * Complete response or partial response: continue at the target dose.
  * No response (stable disease/disease progression):dose reduction to 1/2 dose for 7 days then discontinue treatment.
  Patients who stay on propranolol will undergo tolerability assessments as per the protocol. Patients found to be intolerant of propranolol, or patients who have completed 21 weeks of treatment, will undergo dose reduction to the 1/2 dose for 7 days, and then propranolol will be discontinued.
  Interventions: Drug: Propranolol Hydrochloride

INTERVENTIONS:
Drug: Propranolol Hydrochloride — Dosing is as follows:
  * Patients who weigh 40 to 59.9 kg:
    * 40 mg BID (target)
    * 20 mg BID (half the target)
  * Patients who weigh ≥ 60 kg:
    * 60 mg BID (target)
    * 30 mg BID (half the target)

SUMMARY:
Kaposi sarcoma (KS) lesions are initiated by endothelial cells infected with KS herpesvirus (KSHV), also known as human herpesvirus 8 (HHV-8). Lesion progression is driven by abnormal angiogenesis, chronic inflammation, and uncontrolled cell proliferation. KS remains one of the most commonly diagnosed cancers in many African countries where economic constraints prevent successful treatment in most patients. Treatment outcomes in developed countries are also often unsatisfactory in HIV positive patients despite good virological and immunological responses to antiretroviral therapy. Therefore, identification of new oral, safe treatment options for treatment of KS remains a research priority. Given the known anti-angiogenic properties and based on the treatment response with other benign vascular lesions such as infantile hemangioma, propranolol is a good candidate for the treatment of KS. The hypothesis of this study is that treating patients with Kaposi sarcoma with propranolol will result in an overall response rate (complete response rate plus partial response rate) of at least 45%, and that propranolol will be safe and well tolerated in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven Kaposi Sarcoma that is measurable with a millimeter ruler. Patients presenting for both front-line therapy and subsequent-line therapy will be considered.
* Must have two lesions greater than or equal to 4 mm x 4 mm, or one lesion greater than or equal to 8 mm x 8 mm, that are accessible for 4-mm punch biopsy. The patient must have at least 5 more lesions in addition to the lesion(s) being biopsied.
* At least 18 years of age.
* Weight ≥40 kg
* ECOG performance status ≤ 2
* Meets the appropriate HIV-related criteria:

  * If HIV positive, patient must be on antiretroviral therapy (ART) that conforms to local standards of care for at least 12 weeks. HIV positive patients will not be excluded based on CD4 count or HIV viral load.

    * If on ART 12 to 24 weeks, must show evidence of KS progression requiring further systemic treatment.
    * If on ART for > 24 weeks, must show no evidence of regression in the last 8 weeks.
  * If HIV negative, must not show evidence of improvement in the 12 weeks prior to enrollment.
* Propranolol is US FDA pregnancy category C. For this reason, women of childbearing potential must agree to use adequate contraception prior to study entry, for the duration of study participation, and for one month after completion of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, s/e must inform her treating physician immediately.
* Able to take an oral pill.
* Ability to understand and willingness to sign an IRB approved written informed consent document.

Exclusion Criteria:

* Visceral disease causing functional impairment.
* Urgently clinically indicated for immediate cytotoxic chemotherapy. Patients who have received cytotoxic chemotherapy > 4 weeks prior to screening are eligible.
* Prior or concurrent malignancy whose natural history has the potential to interfere with the safety or efficacy assessment of the investigational regimen. Patients with prior or concurrent malignancy that does NOT meet that definition are eligible for this trial
* Currently taking beta-andrenergic antagonist(s) for other indications. Prior use is allowed if the last dose of the beta-andrenergic antagonist is ≥ 5 half-lives of the agent prior to Day -7.
* Currently receiving concurrent treatment with an anticancer therapy. Patients must not have received any anticancer therapies within 4 weeks prior to receiving the first dose of propranolol.
* Currently receiving any other investigational agents.
* A history of allergic reactions or hypersensitivity attributed to compounds of similar chemical or biologic composition to propranolol.
* History of asthma or current diagnosis of obstructive airway disease such as asthma, COPD, or bronchiolitis.
* History of diabetes mellitus, as defined by any of the following: A random blood glucose value of at least 200 mg/dL in the presence of hyperglycemia symptoms (weight loss, blurry vision, thirst, polyuria), fasting plasma glucose value of at least 126 mg/dL, A1c value of at least 6.5%, or two hour plasma glucose value of at least 200 mg/dL during a 75 g oral glucose tolerance test.
* History of uncompensated heart failure, severe sinus bradycardia, sick sinus syndrome, or heart block greater than first degree.
* History of hypotension (systolic blood pressure <90 mmHg or mean arterial pressure <65 mmHg) or orthostasis (>20 mmHg fall in systolic pressure or >10 mmHg fall in diastolic pressure with standing). (Isolated instances of hypotension may not be exclusionary after discussion with PI.)
* Shortness of breath, hemoptysis, or moderate/severe cough not attributable to causes other than KS.
* Bleeding from the mouth or rectum not attributable to causes other than KS.
* Uncontrolled intercurrent illness including, but not limited to: ongoing clinically significant active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
* Concern for KSHV inflammatory cytokine syndrome.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 21 days of study entry.
* Evidence of chronic hepatitis B virus (HBV) that is detectable on suppressive therapy. Patients with evidence of chronic HBV infection with undetectable HBV viral load on suppressive therapy are eligible. HBV testing not required in the absence of known history of infection.
* History of hepatitis C virus (HCV) infection that has not been cured or that has a detectable viral load. Patients with a history of HCV that has been treated and cured are eligible. Patients with HCV infection who are currently on treatment and have an undetectable HCV viral load are eligible. HCV testing not required in the absence of known history of infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-08-20 (Actual); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Through completion of treatment (estimated to be 22 weeks)
  ORR is defined as the proportion of participants with complete response (CR) or partial response (PR) based on AMC KS Response Criteria.

SECONDARY OUTCOMES:
Incidence of intolerable toxicities and treatment-emergent adverse events (TEAEs) based on CTCAE v 5.0. | From start of treatment through 30 days after completion of treatment (estimated to be 26 weeks)
Time to recurrence or progression among responders overall. | Through completion of follow-up (estimated to be 6 months and 22 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Lee Ratner, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
The data shared will consist of all of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Immediately following publication. No end date.
Access Criteria: Anyone who wishes to access the data for any purpose may be granted access to the data.

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu